CLINICAL TRIAL: NCT03346473
Title: The Double Burden of Malnutrition Among Adolescents: Analysis of Data From the Global School-Based Student Health and Health Behaviour in School-Aged Children Surveys in 57 Low-income and Middle-income Countries
Brief Title: The Double Burden of Malnutrition Among Adolescents in Low-income and Middle-income Countries
Status: Completed | Type: Observational
Sponsor: University of Warwick (Other)
Responsible Party: Principal Investigator, Rishi Caleyachetty, Assistant Professor, University of Warwick
Other Study IDs: WAR2017006203
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Stunting; Thinness; Obese
MeSH Terms: conditions — Growth Disorders; Thinness; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents aged 12-15 years in LMICs: No interventions administered

SUMMARY:
Individual-participant data analysis of the Global School-Based Student Health Survey and Health Behaviour in School-Aged Children surveys in 57 LMICs between 2003-2013.

DETAILED DESCRIPTION:
We used the most recent Global School-Based Student Health Surveys (GSHS) and Health Behaviour in School-Aged Children (HSBC) surveys, with data available on height and weight. The GSHS is a World Health Organisation (WHO) initiative, designed to assess health behaviours of adolescents through cross-sectional school-based surveys, across several countries using similar standardised procedures. The HSBC study are WHO sponsored cross-sectional school-based surveys that uses similar standardised procedures to the GSHS to examine the physical and mental health of adolescents in the WHO European Region and North America.

ELIGIBILITY:
Inclusion Criteria:

* Low-income or middle-income countries with completed Global School-Based Student Health Survey or Health Behaviour in School-Aged Children surveys.
* Adolescents aged 12-15 years
* Recorded sex, height and weight

Exclusion Criteria:

- High-income countries

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents aged 12-15 years from the Global School-Based Student Health Surveys (GSHS) and Health Behaviour in School-Aged Children (HSBC) surveys.
Sampling Method: Probability Sample
Enrollment: 129276 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of stunting | 2003-2013
  Trained survey staff measured the height of each student. Stunting was defined as height-for age < 2 standard deviations below the WHO Child Growth Reference median.
Prevalence of thinness | 2003-2013
  Trained survey staff measured the weight of each student. Thinness was defined as BMI-for-age < 2 standard deviations below the WHO Growth Reference median. Body mass index [BMI (weight in kilograms divided by height in meters squared)] was calculated from height and weight.
Prevalence of overweight and obesity | 2003-2013
  Overweight was defined as BMI-for-age > 1 standard deviation above the WHO Growth Reference median) and obesity was defined as >2 standard deviations above the WHO Growth Reference median.

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Caleyachetty, MBBS PhD, Principal Investigator — Warwick Medical School, Warwick University

REFERENCES:
- [Derived] Caleyachetty R, Thomas GN, Kengne AP, Echouffo-Tcheugui JB, Schilsky S, Khodabocus J, Uauy R. The double burden of malnutrition among adolescents: analysis of data from the Global School-Based Student Health and Health Behavior in School-Aged Children surveys in 57 low- and middle-income countries. Am J Clin Nutr. 2018 Aug 1;108(2):414-424. doi: 10.1093/ajcn/nqy105. PMID 29947727